CLINICAL TRIAL: NCT04097093
Title: Long-term Survival of Advanced/Metastatic GIST Patients Responding to Imatinib Treatment: an Observational Follow-up Study
Brief Title: Long-term Surival of GIST Patients ≥ 10 Years on Imatinib
Status: Withdrawn | Type: Observational
Why Stopped: Lack of feasibility
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC 1826-STBSG
Record Dates: First submitted 2019-08-07; First posted 2019-09-20 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: GIST

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — First, existing data on molecular characteristics of included patients will be collected from the treating centers. If more than 40% of the data is not available, archival tumor tissue from patients enrolled in the EORTC 62005-STBSG study will be collected and used to identify molecular characteristics of the tumor that may predict long-term response to imatinib. Archival tumor tissues will be retrieved from the central lab of the study 62005-STBSG (UZ Leuven, Belgium) or from the sites (if applicable).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study 62005-STBSG patients treated with imatinib > 10 years
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a cross-sectional cohort study of metastatic GastroIntestinal Stromal Tumor (GIST) patients on imatinib for ≥ 10 years included in EORTC trial 62005-STBSG entitled "Phase 3 randomized, intergroup, international tiral assessing the clinical activity of STI-571 at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumor (GIST) expressing the KIT receptor tyrosine kinase (CD117) - NCT00685828". With this study, the aim is to identify patient characteristics, tumour characteristics, treatment factors and quality of life outcomes associated with prolonged treatment with imatinib and/or prolonged survival. This observational study will further help to put in place a questionnaire to evaluate patients quality of life with prolonged imatinib treatment, that will then be used in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the EORTC 62005 trial: Adult patients with metastasized GIST
* Patients who have been treated with imatinib for ten years or longer
* For the identified patients who are still alive:

  1. Able to read and answer questionnaires
  2. Able to provide written informed consent

Min Age: 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the 62005 trial - treated for more than 10 years with imatinib - will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics | At time of registration
  Age at time of randomization, gender, medical history and previous treatment(s)
Tumour characteristics | At time of registration
  Stage of the disease, tumor grade, tumor location and molecular features of primary tumor
Duration of imatinib treatment | At time of registration
  Time on imatinib treatment from start untill definitive discontinuation of imatinib treatment
Health releated quality of life | At time of registration
  QLQ-C30
Overall survival | At time of registration
  From time of randomization to the date of death, whatever the cause

CONTACTS AND LOCATIONS:
Overall Officials: Neeltje Steeghs, Study Chair — NKI - Antoni van Leeuwenhoekziekenhuis; Axel Le Cesne, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Ingrid Desar, Study Chair — Radboud University Medical Center Nijmegen; Olga Husson, Study Chair — Radboud University Medical Center Nijmegen

IPD SHARING:
Plan to Share IPD: No